CLINICAL TRIAL: NCT04890886
Title: Magnetic Resonance Imaging and Thermal Imaging of Adiposity in Neonates of Women With Metabolic Diseases
Acronym: MRI-TIME
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 287911
Record Dates: First submitted 2021-05-13; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Diabetes Mellitus; Intrahepatic Cholestasis of Pregnancy; Metabolic Disease
Keywords: type 1 diabetes; type 2 diabetes; gestational diabetes; intrahepatic cholestasis of pregnancy; metabolic disease in pregnancy; brown adipose tissue; white adipose tissue; cardiac function; ECG; liver function; thermal imaging
MeSH Terms: conditions — Diabetes Mellitus; Intrahepatic Cholestasis of Pregnancy; Metabolic Diseases; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes, Gestational | interventions — Echocardiography; Electrocardiography; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples to measure metabolic function and measures of cardiac function
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pre-existing Type 1 Diabetes and Type 2 Diabetes: Women with type 1 diabetes and type 2 diabetes diagnosed prior to pregnancy
  Interventions: Diagnostic Test: Thermal imaging; Diagnostic Test: Echocardiogram; Diagnostic Test: ECG; Diagnostic Test: MRI scan; Diagnostic Test: Serum blood markers
- Gestational Diabetes: Women with gestational diabetes diagnosed in pregnancy by the oral glucose tolerance test
  Interventions: Diagnostic Test: Thermal imaging; Diagnostic Test: Echocardiogram; Diagnostic Test: ECG; Diagnostic Test: MRI scan; Diagnostic Test: Serum blood markers
- Intrahepatic cholestasis of pregnancy: Women with intrahepatic cholestasis of pregnancy
  Interventions: Diagnostic Test: Thermal imaging; Diagnostic Test: Echocardiogram; Diagnostic Test: ECG; Diagnostic Test: MRI scan; Diagnostic Test: Serum blood markers
- Control: Women without metabolic disease in pregnancy
  Interventions: Diagnostic Test: Thermal imaging; Diagnostic Test: Echocardiogram; Diagnostic Test: ECG; Diagnostic Test: MRI scan; Diagnostic Test: Serum blood markers

INTERVENTIONS:
Diagnostic Test: Thermal imaging — Use of a thermal imaging cameral to measure brown and white adipose tissue function
Diagnostic Test: Echocardiogram — Echocardiographic imaging of the fetal heart to assess ventricular function
Diagnostic Test: ECG — ECG of the fetus and the neonate to look at the cardiac electrical activity
Diagnostic Test: MRI scan — MRI scan of the neonate to assess adipose tissue, liver architecture and cardiac structure and function
Diagnostic Test: Serum blood markers — Serum sample taken from mother before birth and umbilical cord or neonatal blood spot at birth to assess glucose levels / lipid levels and lipidomics and cardiac function (using NTproBNP) as a marker

SUMMARY:
There is limited knowledge about the extent of the impact of maternal metabolic diseases (MD) and/or alterations in maternal serum lipid content upon neonatal lipid distribution and phenotypes. This observational feasibility study aims to investigate the effect of maternal MD on fat distribution, lipid content and metabolic phenotype of different neonatal tissues. We will explore whether differences in tissue fat distribution and lipid content are observed in the neonates of women with MD during pregnancy, compared to those who have a healthy, uncomplicated pregnancy and if there are changes in how the different tissues work (e.g. cardiac function). If there is evidence to show that there are alterations during pregnancy in children of women with MD, this will help inform potential interventions to ensure optimal child health.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women aged between 16 and 45 years old.
2. Women with GDM diagnosed at 26+0 to 30+6 weeks' gestation in accordance with the NICE guidelines Or
3. Pregnant women with pre-existing type 1 or type 2 diabetes mellitus Or
4. Women diagnosed with ICP at any stage of pregnancy
5. Fluent in English or presence of an interpreter or translation service (i.e. telephone translation services) at all visits.
6. Singleton pregnancy.
7. Willing and able to give written informed consent and comply with requirements of the study protocol
8. Planned antenatal, intrapartum and postpartum care at the participating centre (i.e. not planning to move before delivery)

Exclusion Criteria:

1. Known fetal congenital abnormality on ultrasound requiring fetal medicine input (excluding congenital heart disease).

1. Known fetal congenital abnormality on ultrasound requiring fetal medicine input (excluding congenital heart disease).
2. Significant pre-pregnancy co-morbidities that increase risk in pregnancy, for example renal failure, severe liver disease, transplantation, cardiac failure, psychiatric conditions requiring in-patient admission (within previous year) in the opinion of the responsible clinician or the CI.
3. Significant co-morbidity in the current pregnancy, nephropathy (estimated GFR <60ml/min), other physical or psychological conditions likely to interfere with the conduct of the study and/or interpretation of the study results in the opinion of the responsible clinician or the CI. (This does not include diabetes mellitus).
4. History of bariatric surgery.
5. Hypertension requiring treatment pre-pregnancy / in pregnancy.
6. Prescribed other medications that affect insulin sensitivity prior to OGTT for women diagnosed with GDM (oral antihyperglycemic agents, antipsychotic drugs, supraphysiological doses of steroids).
7. For the baby after birth: Not meeting the safety criteria to undergo MRI scan (e.g. metal implants, non MRI compatible devices, metal fragments in the body). [ The mother will not have an MRI scan].

Ages: 16 Years to 45 Years | Sex: Female
Age Groups: Child, Adult
Study Population: Pregnant women with metabolic disease in pregnancy or healthy controls.
  The neonates that will be studied can be of any sex/gender for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the distribution of adipose tissue | 30 months
  To perform imaging and biochemical studies to determine whether maternal metabolic disease alters the distribution of adipose tissue (SAT, VAT, BAT) of the fetuses and neonates of women with MD during pregnancy compared to neonates of women who had a healthy pregnancy.

SECONDARY OUTCOMES:
Assessment of skeletal muscle, heart and liver | 30 months
  To perform imaging and biochemical studies to determine whether maternal metabolic disease alters the distribution and phenotypes of skeletal muscle, heart and liver of the fetuses and neonates of women with MD during pregnancy compared to those of women who had a healthy pregnancy.
Assessment of the function of adipose tissue | 30 months
  To evaluate novel MRI-based techniques to measure the function of adipose tissue (SAT, VAT, BAT) in the neonates.
Assessment of cardiac function and rhythm | 30 months
  To perform echocardiography and fetal/ neonatal ECG studies to understand the impact of maternal MD on the fetal heart.
Thermal assessment | 30 months
  To use thermal imaging to determine the temperature of regions of interest, e.g. BAT, of pregnant women with MD and their neonates.

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be made available upon reasonable request and final decision from the PI.